CLINICAL TRIAL: NCT02645500
Title: The Efficacy of Training Programme and Mobile Health Message on Promoting Family Holistic Health
Brief Title: Training Program and Mobile Health Message on Promoting Family Holistic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Research Officer, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW15-478
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity; Health Behavior; Quality of Life
Keywords: Physical Activity; Family well-being
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity message (Experimental): Participants will receive training on healthy living style focusing on positive psychology, physical activity and healthy diet, and health messages related to physical activity.
  The training workshop include one core session and one booster session at one month.
  Daily messages in relation to physical activity will be sent to the participants.
  Interventions: Behavioral: Holistic health training and physical exercise messages
- Healthy diet message (Active Comparator): Participants will receive training on healthy living style focusing on positive psychology, physical activity and healthy diet, and health messages related to healthy diet .
  The training workshop include one core session and one booster session at one month.
  Daily messages in relation to healthy diet will be sent to the participants.
  Interventions: Behavioral: Holistic Health Training with healthy diet messages

INTERVENTIONS:
Behavioral: Holistic health training and physical exercise messages — The physical activity message arm includes a training workshop in relation to holistic health, and daily physical activity messages.
  Arms: Physical activity message
Behavioral: Holistic Health Training with healthy diet messages — The healthy diet message arm includes a training workshop in relation to holistic health, and daily healthy diet messages.
  Arms: Healthy diet message

SUMMARY:
In this study, the investigators would use the training workshops as a capacity build method to deliver the holistic health knowledge for the trainers and ambassadors implementing and assisting the community-based programs for the public. The investigators hypothesize that the training workshops and mobile health messages would promote the health awareness and the health of the participants. The investigators would expect the participants influence the health behavior and attitude of their family members.

DETAILED DESCRIPTION:
Holistic health is an integration and interaction of physical and psychosocial health. Positive psychology is a science of happiness, which focuses on positive emotions and personal strengths. It is used as a preventive and complementary medicine, which also is crucial component in family holistic health (happiness, harmony and health). Healthy diet can help to achieve energy balance and healthy weights. Sufficient daily consumption of fruit and vegetables, as well as limitation on the intake of sugar, salt and fat could prevent major diseases, such as cardiovascular diseases and certain cancers. Physical activity is believed to contribute to physical and mental health, as well as social well-being. However, physical inactivity was found to be a local and worldwide issue. and most Hong Kong people are having sedentary lifestyle. Studies show that the increase of physical activity and healthy diet reduce the risk of chronic diseases, and improve cardio-pulmonary functions; whereas sedentary behaviors increase the risk.

The Project team will schedule the training workshops for the trainers and ambassadors implementing and assisting community-based programs for the public. The investigators hypothesize that the training workshops and mobile health messages would promote the health awareness and the health of the participants. The investigators hypothesize that the training workshops promote the participants' knowledge and enhance the participants' behaviors related to family holistic health, such as positive psychology, physical activity and healthy diet. The investigators would expect the participants influence the health attitude of their family members.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking
* able to complete study questionnaire

Exclusion Criteria:

* not fit the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge in relation to physical activity | Baseline and one month
  Change in knowledge in relation to physical activity will be assessed by outcome-based questionnaire (a visual analogue scale)

SECONDARY OUTCOMES:
Change in knowledge in relation to physical activity | Baseline, immediately after core session, one month, and three months
  Change in knowledge in relation to physical activity will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in attitude on performing physical activity | Baseline, immediately after core session, one month, and three months
  Change in attitude on performing physical activity will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in health behaviour in relation to physical activity | Baseline, immediately after core session, one month, and three months
  Change in health behaviour on performing physical activity will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in quality of life | Baseline, one month and three months
  Change in quality of life will be assessed by SF12 v2 health survey (a visual analogue scale)
Change in personal happiness | Baseline, one month and three months
  Change in subjective happiness will be assessed by outcome-based questionnaire ( a visual analogue scale)
Change in personal health | Baseline, one month and three months
  Change in personal health will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in family well-being | Baseline, one month and three months
  Change in family well-being will be assessed by family well-being scale (a visual analogue scale)
Change in knowledge sharing with family members in relation of physical activity | Baseline, one month, three months
  Change in knowledge sharing with family members in relation to physical activity will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in knowledge sharing with family members in relation of healthy diet | Baseline, one month, three months
  Change in knowledge sharing with family members in relation to healthy diet will be assessed by outcome-based questionnaire ( a visual analogue scale)
Change in behavior to appraise family members | Baseline, one month, three months
  Change in behavior to appraise family members will be assessed by outcome-based questionnaire ( a visual analogue scale)
Change in health behavior of performing physical activity with family members | Baseline, one month, three months
  Change in health behavior of performing physical activity with family members will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in health behavior of taking healthy diet with family members | Baseline, one month, three months
  Change in health behavior of taking healthy diet with family members will be assessed by outcome-based questionnaire (a visual analogue scale)
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Balance will be assessed through a simple fitness test called single-leg stand (measuring seconds).
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Muscle endurance will be assessed through a simple test called Chair-to-stand ( measuring unit: time).
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Flexibility will be assessed through a simple fitness test called seat and reach (measuring unit: cm).
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Body mass index will be assessed through body weight and body height measuring scales (measuring unit: BMI in kg/m^2, weight in kilograms, height in meters) .
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Lower limb muscle strength will be assessed through a vertical jump measuring device (measuring unit: cm ).
Change in physical fitness | Baseline, one month
  Physical fitness will be assessed by simple physical tests. Handgrip strength will be assessed through handgrip dynamometers (measuring unit: kg) .
Satisfaction towards training program | immediately after core session, immediately after one-month booster session
  Satisfaction towards training session will be assessed by a program evaluation outcome-based questionnaire ( a visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, DN, Principal Investigator — The University of Hong Kong
Locations (1):
- The Boys' and girls' association of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshikawa H. Integrating methods in the science of family health: new directions from an institute of medicine workshop report. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):659-61. doi: 10.1001/archpediatrics.2012.510. No abstract available. PMID 22751883
- [Background] Bellicha A, Kieusseian A, Fontvieille AM, Tataranni A, Charreire H, Oppert JM. Stair-use interventions in worksites and public settings - a systematic review of effectiveness and external validity. Prev Med. 2015 Jan;70:3-13. doi: 10.1016/j.ypmed.2014.11.001. Epub 2014 Nov 10. PMID 25449692
- [Background] Radtke T, Rackow P. Autonomous motivation is not enough: the role of compensatory health beliefs for the readiness to change stair and elevator use. Int J Environ Res Public Health. 2014 Nov 28;11(12):12412-28. doi: 10.3390/ijerph111212412. PMID 25464134
- See also: Department of Health: Physical activity — http://www.dh.gov.hk/english/useful/useful_dykt/useful_dykt_exercise.html